CLINICAL TRIAL: NCT00711711
Title: Outcome of Manual Lymphatic Drainage Following Total Knee Arthroplasty Surgery
Brief Title: Manual Lymphatic Drainage Following Total Knee Arthroplasty Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Haute Ecole de Santé Vaud (Other)
Collaborators: University of Applied Sciences of Western Switzerland (Other); University of Lausanne Hospitals (Other)
Responsible Party: Principal Investigator, Claude Pichonnaz, Associate professor, Haute Ecole de Santé Vaud
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: FNS-DORE 13DPD3-120298; SAGEX: 21267 (Other: HES-SO); RéSaR 10/O/07 (Other: HES-SO); Ré-Sa-R 13-07 (Other: HES-SO)
Record Dates: First submitted 2008-07-08; First posted 2008-07-09 (Estimated); Results first posted 2019-01-18 (Actual); Last update posted 2019-01-18 (Actual); Status verified 2018-08

CONDITIONS: Knee Arthroplasty, Total
Keywords: Physical Therapy - Therapeutics - Edema; Arthroplasty replacement knee; Treatment outcome
MeSH Terms: interventions — Manual Lymphatic Drainage

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Manual lymphatic drainage (Experimental): this arm will receive 5 manual lymphatic drainage treatments from day 2 to day 7 post surgery
  Interventions: Other: Manual lymphatic drainage
- Relaxation (Placebo Comparator): This arm will receive 5 relaxation treatments from day 2 to day 7 post surgery
  Interventions: Other: relaxation

INTERVENTIONS:
Other: Manual lymphatic drainage — Each patient will receive 5 treatments of 30 minutes by a trained physiotherapist, from day 2 to day 7 post surgery
  Other Names: lymphatic drainage; manual lymph drainage; MLD
  Arms: Manual lymphatic drainage
Other: relaxation — Each patient will receive 5 treatments of 30 minutes of tape recorded relaxation , from day 2 to day 7 post surgery
  Other Names: eriksonian hypnosis
  Arms: Relaxation

SUMMARY:
The purpose of this study is to evaluate the efficiency of manual lymphatic drainage to decrease the swelling of the knee after total knee replacement surgery

DETAILED DESCRIPTION:
Background There is scientific evidence that rehabilitation has a positive influence on patients'recovery after total knee arthroplasty (TKA). According to the literature, conventional rehabilitation aims to improve knee range of motion, lower limb strength, gait, activities and pain. Although swelling is a systematic consequence of TKA surgery, less focus is put on swelling reduction. Patients develop swelling due to periarticular edema, hematoma and joint effusion. Inflammation, pain, stiffness, alteration of gait pattern, quadriceps contraction inhibition and slowing of rehabilitation are reported as consequences of swelling. Accordingly, it is likely that a therapy that would promote resorption of swelling would decrease the negative impact of swelling on patients'recovery. Manual lymph drainage (MLD) could possibly accelerate edema resorption after TKA surgery. Several authors advise MLD after TKA, and physiotherapists currently apply MLD to reduce postsurgical swelling. Its positive effect on chronic lymphedema resorption is largely accepted. Results on pain and range of motion seem interesting from an empirical point of view but, to our knowledge, no scientifically driven studies have confirmed these positive effects after orthopaedic surgery.

Aim This study aims to evaluate the effect of MLD on swelling, and parameters possibly influenced by swelling (pain, knee range of motion, knee objective and subjective function and gait pattern).

Methods This study is a randomized controlled clinical trial. Patients will be blinded from goals of the treatments and evaluators will be blinded from the treatment delivered to the patient. The effects of MLD (5 treatments of 30 minutes from the second to the eighth postsurgical day) will be compared to those of a placebo (relaxation sessions). MLD or placebo will be added to the conventional rehabilitation program of our Orthopaedic Department. Assessments will be conducted one day before surgery, two days, 8 days and 3 months after surgery. Evolution and differences between groups will be statistically assessed at each step.

Significance This project aims to improve knowledge on the efficiency of rehabilitation treatments following TKA. It will contribute to effective evaluation of the effects of a widely applied treatment. The results will help physiotherapists and medical doctors to take clinical decisions based on documented evidence. This will make a contribution to better quality of care and better allocation of resources to rehabilitation.

ELIGIBILITY:
Inclusion Criteria:

* knee replacement surgery

Exclusion Criteria:

* pacemaker
* cardiac defibrillator
* pathology of the lymphatic system
* lower limb impairment which interferes with gait
* neurological disease
* unability to understand patient information letter or to give informed consent
* unability to understand and complete questionnaires in French
* contraindication to manual lymphatic drainage : thrombosis, infection, right cardiac insufficiency, active cancer
* non standard knee replacement surgery
* high dose anticoagulation
* post surgical complication

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2008-06; Primary Completion 2011-01 (Actual); Study Completion 2011-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Claude Pichonnaz, physiother, Principal Investigator — Haute Ecole Cantonale Vaudoise de Santé + Département de l'Appareil Locomoteur - CHUV; Brigitte M Jolles, PD MER MSc, Study Director — Département de l'Appareil Locomoteur - CHUV + Faculté des sciences et techniques de l'ingénieur (STI) - EPFL
Locations (2):
- Switzerland (2):
  - Département de l'Appareil Locomoteur - CHUV, Lausanne
  - Haute Ecole Cantonale Vaudoise de Santé, Lausanne

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pichonnaz C, Bassin JP, Lecureux E, Christe G, Currat D, Aminian K, Jolles BM. Effect of Manual Lymphatic Drainage After Total Knee Arthroplasty: A Randomized Controlled Trial. Arch Phys Med Rehabil. 2016 May;97(5):674-82. doi: 10.1016/j.apmr.2016.01.006. Epub 2016 Jan 30. PMID 26829760

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients from the Department of Orthopedic and Traumatic Surgery of the University Hospital of Lausanne were recruited from July 1, 2008 to November 16, 2010
Period: Overall Study
Arm/Group | Manual Lymphatic Drainage | Relaxation
Started | 30 | 30
Second Postsurgical Day | 30 | 30
Seventh Postsurgical Day | 29 | 27
Completed | 29 | 24
Not Completed | 1 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Manual Lymphatic Drainage | Relaxation | Total
Number analyzed (Participants) | 30 | 30 | 60
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 23 | 21 | 44
  >=65 years | 7 | 9 | 16
Age, Continuous [Mean (Standard Deviation); unit: years] | 71.3 (8.5) | 70.1 (9.1) | 70.7 (8.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 21 | 39
  Male | 12 | 9 | 21
Region of Enrollment [Number; unit: participants]
  Switzerland | 30 | 30 | 60

OUTCOME MEASURES:

1. Primary Outcome: Bioimpedance Percentage Difference Healthy/Operated
Description: The bioimpedance, i.e. a measurement in ohms of the opposition to current flow between electrodes was evaluated for each limb. Then the bioimpedance percentage difference between operated and healthy limb was calculated.
Time Frame: presurgery, 2 days, 7 days and 3 months post surgery
Population: At day 7, 3 patients lost at follow up in the control group and 1 in the treatment group.
  At 3 months, 3 more patients lost at follow up in the control group.
Measure: Mean (Standard Deviation); unit: percentage difference between limbs
Groups:
- Placebo: Patients who received relaxation as placebo intervention
- Manual Lymphatic Drainage: Patients who received manual lymphatic drainage as the study intervention
Arm/Group | Placebo | Manual Lymphatic Drainage
Number analyzed (Participants) | 30 | 30
percentage difference between limbs
  Baseline limb bioimpedance R0 difference (%) | 1.8 (5.0) | 0.2 (4.5)
  Limb bioimpedance R0 difference at day 2 (%) | 12.9 (9.7) | 13.7 (72)
  Limb bioimpedance R0 difference at day 7 (%): number analyzed (Participants) | 27 | 29
  Limb bioimpedance R0 difference at day 7 (%) | 41.8 (6.5) | 40.8 (6.6)
  Limb bioimpedance R0 difference at 3 months (%): number analyzed (Participants) | 24 | 29
  Limb bioimpedance R0 difference at 3 months (%) | 16.6 (9.3) | 19.1 (11.0)
Statistical Analysis 1: Comparison: Placebo vs Manual Lymphatic Drainage; All outcomes and control variables were compared between the treatment and the control group at each time point using the Wilcoxon rank-sum test or the chi-square test, as appropriate. The change in swelling from second day to seventh day, that is, during the treatment period, was compared using the Wilcoxon signed-rank test. The significance level was set at P<.05; Test type: Superiority or Other; p = 0.51, Wilcoxon (Mann-Whitney)

2. Primary Outcome: Lower Limb Volume Percentage Difference Operated/Healthy
Description: The limb volume was evaluated for each limb using circumferential tape measurements at 4 cm intervals. Then the tape measurementy were converted into limb volume using the validated truncated-cone method, and the percentage difference between the operated and the healthy limb was calculated.
Time Frame: presurgery, and 2 days, 7 days and 3 months after surgery
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage difference between limbs
Arm/Group | Manual Lymphatic Drainage | Relaxation
Number analyzed (Participants) | 30 | 30
percentage difference between limbs
  Baseline limb volume difference (%) | 1.8 (5.0) | 0. (4.5)
  Limb volume difference at day 2 (%) | 12.9 (9.7) | 13.7 (7.2)
  Limb volume difference at day 7 (%): number analyzed (Participants) | 29 | 27
  Limb volume difference at day 7 (%) | 17.0 (10.7) | 15.3 (6.5)
  Limb volume difference at 3 months (%): number analyzed (Participants) | 29 | 24
  Limb volume difference at 3 months (%) | 3.7 (5.7) | 4.1 (5.1)
Statistical Analysis 1: Comparison: Manual Lymphatic Drainage vs Relaxation; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.58, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Arm/Group | Manual Lymphatic Drainage | Relaxation
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/30
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30
Other Adverse Events (participants affected / at risk) | 0/30 | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes